CLINICAL TRIAL: NCT02893774
Title: Longitudinal Study of Behavioral Changes, Economic and Sociological After CAncer
Acronym: ELCCA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2014-10; 2014-A01675-42 (Other: ANSM)
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Melanoma
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cancer quality of life (Experimental): All patients with breath cancer or melanoma will have quality of life assessment 1, 6, 12, 24, 48 and 60 months after the initial cancer diagnosis
  Interventions: Other: quality of life assessment

INTERVENTIONS:
Other: quality of life assessment — All patients with breath cancer or melanoma will have quality of life assessment 1, 6, 12, 24, 48 and 60 months after the initial cancer diagnosis.
  Those assessment will use standardized quality of life questionnaire :
  * QLQ-C30
  * SWLS (Satisfaction with Life Scale)
  * PTGI (Post-Traumatic Growth Inventory)
  * HADS (Hospital Anxiety and Depression Scale)
  * Brief COPE
  * MHLCS (Multidimensional Health Locus of Control Scale)

SUMMARY:
Generally, French studies concerned with the quality of life of cancer patients focus on the period of treatment (up to 2 years post diagnosis). However, studies about quality of life "after" cancer are relatively rare (= long-term quality of life, or from 5 years post diagnosis). These studies mainly concern the most common cancers (breast and prostate).

Or changes in quality of life after treatment could be different depending on the type of cancer. In addition, there is a significant influence of sociodemographic variables on the quality of life in remission.

Similarly using remote diagnostics, quality of life questionnaires related to health, must be reassessed because too often developed for situations in process.

Based on these findings, "ELCCA II" study proposes to study for five years, the evolution of the impacts of two types of cancer (breast and melanoma) on quality of life (overall and related to the subjective health), socioeconomic status, and behavioral and emotional dimensions (post-traumatic development, coping, anxiety-depression) of those treated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer (breast or melanoma) since less than 1 month
* no metastasis
* Inform Consent Form signed

Exclusion Criteria:

* severe psychiatric disorder (depression, psychosis, etc.)
* addictive pathology
* longtime antidepressant treatment (> 3 months)
* Patient pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
long term evolution of quality of life for patient with breast cancer or melanoma | 5 years after initial cancer diagnostics
  The evolution of quality of life will be assess with standardized quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: CAMPONE Mario, Pr, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO René Gauducheau, Nantes, France

IPD SHARING:
Plan to Share IPD: No